CLINICAL TRIAL: NCT02033109
Title: A Phase 1, Double-Blind, Parallel, Placebo-Controlled, Randomized Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Acceptability of PC-1005 Microbicide Gel Formulation in HIV-seronegative Women
Brief Title: Safety, Pharmacokinetics and Acceptability of PC-1005 for Vaginal Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Population Council #558
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PC-1005 (Experimental): * 4.00 g dosed once daily for 3 days (safety run-in)
  * 4.00 g dosed once daily for 14 days (main study)
  Interventions: Drug: PC-1005
- HEC gel (Placebo Comparator): 4.00 g dosed once daily for 14 days (main study only)
  Interventions: Drug: HEC gel

INTERVENTIONS:
Drug: PC-1005 — Intravaginal use
  Other Names: MIV-150/zinc acetate in a carrageenan gel
  Arms: PC-1005
Drug: HEC gel
  Other Names: hydroxyethylcellulose gel; placebo gel
  Arms: HEC gel

SUMMARY:
This Phase 1 clinical trial will evaluate MIV-150, a third generation non-nucleoside reverse transcriptase inhibitor, co-formulated with a potentially potent agent, zinc acetate for the prevention of HIV infection in women. This is the first in-human of PC-1005 (MIV-150/zinc acetate in a carrageenan gel), the first study in which females will be exposed to MIV-150, the first time MIV-150 will be administered topically, and the first time MIV-150 will be administered intravaginally.

DETAILED DESCRIPTION:
This study will begin with a safety run-in, which is an open label, single-arm safety run-in with 5 women receiving PC-1005 once daily for 3 consecutive days. Safety and pharmacokinetics will take place after each dose. the participants from the run-in will not be eligible for the main study.

The main study participants will be randomized 4:1 to the study gels: 24 randomized to PC-1005 (active) and 6 randomized to HEC gel (placebo). The study product will be applied vaginally once daily for 14 days with clinical and laboratory assessments at baseline (enrollment) and after the 1st, 2nd, 8th, 9th, and 14th doses, and a safety follow-up visit 7 days after the 14th dose.

Participants in the run-in and main study will be requested to be sexually abstinent starting immediately after the Screening Visit until study exit.

ELIGIBILITY:
Inclusion Criteria:

* Women between 19 and 49 years of age, inclusive
* Willing and able to provide written informed consent
* Healthy, based on medical history, vital signs, physical examination, urinalysis, laboratory evaluations for genital infections and laboratory evaluations for hematology, liver and renal function with a BMI ≥18 kg/m^2 and ≤32 kg/m^2
* HIV-negative as determined by HIV ELISA test at screening
* Hepatitis B and C negative at screening
* Rapid plasma reagin negative at screening
* If HSV-2 positive, must be free from outbreaks for at least 6 months prior to screening
* In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle, defined as having a minimum of 21 days and a maximum of 35 days between menses
* Normal Pap test at screening
* Agrees to use one form of effective contraception for the duration of the trial
* Willing to abstain from sexual intercourse/activity including receptive vaginal, oral, digital, and anal intercourse, and the use of any vaginal products including tampons, male and female condoms, contraceptive sponges, diaphragms, cervical caps, douches, lubricants, and vibrators/dildos starting from the Screening Visit through Study Exit
* Agrees to not participate in any other clinical research trial for the duration of this trial

Exclusion Criteria:

* History of or known sensitivity/allergy to any component of either study product
* Currently pregnant or breast-feeding, or within 3 months of last pregnancy outcome
* Participation in any other clinical research trial involving investigational or marketed products currently or within two months of participation prior to screening, including any trial of a spermicide, microbicide and/or drug
* Diagnosed with or treated for any STI (other than HSV) or pelvic inflammatory disease in the last 3 months
* Positive test for Neisseria gonorrhea, Chlamydia trachomatis, or Trichomonas vaginalis
* Symptomatic vulvovaginal candidiasis, bacterial vaginosis (BV), or urinary tract infection (UTI) at screening
* Presence of any clinically significant genital epithelial findings such as abrasions, ulcerations, lacerations, or vesicles suspicious for STIs at screening
* Presence of any other clinically significant abnormal physical finding on the vulva, vaginal walls or cervix at screening
* Any clinically significant abnormal hematology, chemistry or urinalysis findings at screening
* Any chronic (excluding HSV-2) or progressive disease (including any known history of cancer, diabetes, cardiac disease, autoimmune disease, blood dyscrasias, or Wilson's disease), or signs of cardiovascular disease, or renal failure, even controlled with medication
* History of hysterectomy or menopause
* Use of excluded contraceptive methods including Nuvaring®, condoms (male or female), contraceptive sponge, diaphragm, or cervical cap (Safety Run-in and Main study)
* History of gynecological surgery or procedure within past 2 months
* History of uterine prolapse, undiagnosed vaginal bleeding or urethral obstruction within the last 3 months, including break-through bleeding requiring sanitary protection
* Known current drug abuse, including illicit drugs, or alcohol abuse
* Any other condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives
* Unable to comply with study requirements, including but not limited to, attending all study visits, using the gel as directed, observing abstinence throughout the study and use of effective contraceptives, limiting alcoholic beverages to 2 per day and caffeine to no more than 6 servings per day
* History of latex allergy

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety: adverse events, serious adverse events, physical exams, and clinical laboratory parameters | 5 weeks for safety run-in study; 7 weeks for main study
  * Number and percent of participants with treatment emergent adverse events and adverse events, and medical significance of adverse events and serious adverse events
  * Number, percent and medical significance of abnormalities in physical exams, pelvic exams, and biopsies once product has been administered
  * Number, percent and medical significance of abnormalities in clinical laboratory parameters once product has been administered

SECONDARY OUTCOMES:
Assessment of acceptability and adherence of PC-1005 use in seronegative women (main study only) | 14 days
  Questionnaire, self-report, and applicators returned empty

OTHER OUTCOMES:
Exploratory: pharmacodynamics and immune mediators | Day 1 (baseline, both run-in and main); Day 14 (post-dose, main study only)
  * Anti-HIV, anti-HSV, and anti-HPV activity in cervicovaginal lavages (CVL)
  * Immune mediators in CVL
Exploratory: MIV-150 and zinc levels in cervical tissue biopsies (main study only) | Day 14 (post-dose)
  Additional cervical biopsy after the last dose
Exploratory: dye stain assay analysis | Post-dose
  * Sensitivity, specificity, negative predictive values and positive predictive values of the dye stain assay, using applicators inserted under direct observation as the positive controls
  * Correlation between self-reported adherence, pharmacokinetics, pharmacodynamics, number of returned applicators and dye stain assay
Exploratory: pharmacokinetics evaluation of zinc in resum | Days 1, 2 and 3 (run-in) / Days 1, 8 and 14 (main study)

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Hoesley, MD, Principal Investigator — University of Alabama at Birmingham; George W Creasy, MD, Study Chair — Population Council; Barbara Friedland, MPH, Study Director — Population Council
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States